CLINICAL TRIAL: NCT01331759
Title: Neuropattern™ Stress Diagnostics in Workplace Health Promotion
Brief Title: Neuropattern™ for Workplace Health Promotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daacro (Network)
Collaborators: University of Trier (Other)
Responsible Party: Principal Investigator, Juliane Hellhammer, MSc, Daacro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LF1-2010
Record Dates: First submitted 2011-04-01; First posted 2011-04-08 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Stress-Related Disorder
Keywords: Burnout; Subthreshold Disorder
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Neuropattern™ (Experimental): The experimental group will undergo Neuropattern™ stress diagnostics immediately after inclusion in the study.
  Interventions: Device: Neuropattern™
- Later Neuropattern™ (Placebo Comparator): The control group will undergo Neuropattern™ stress diagnostics three months after inclusion in the study.
  Interventions: Device: Neuropattern™

INTERVENTIONS:
Device: Neuropattern™ — Neuropattern™ is a diagnostic tool aiming at measuring states of activity and reactivity of interfaces involved in the communication between the brain and peripheral bodily organs in stressful situations. The concept of Neuropattern™ assumes the states of the various interfaces to be describable by characteristic patterns of simultaneous activation of biological, psychological and symptomatic variables. Neuropattern™ assesses endophenotypes through the medical history, various questionnaires for the patient or study subject, analyses of saliva cortisol and the heart rate variability and derives hypotheses on recommendations for an effective and efficient treatment.These recommendations are based on evaluated medical and psychological therapeutic methods but specified through additional biopsychological understanding. This form of individualized therapy should reduce nonresponsiveness to therapy.
  Other Names: Stress Diagnostics; Translational Medicine

SUMMARY:
Neuropattern™, a new diagnostic tool for stress related disorders is being applied in a demanding workplace environment. Neuropattern™ aims at identifying stress-related bodily changes at an early stage. By identifying subgroups based on Neuropattern™ subjects gain access to online counseling specified according to their Neuropattern™ diagnosis. Efficacy is being assessed by several questionnaires in a follow-up.

DETAILED DESCRIPTION:
100 employees of a company in Rhineland Palatinate employing approximately 2100 persons will be recruited.

This is a randomized, two-armed single center study. Persons interested in study participation receive a Neuropattern™ voucher according to occupational group together with other documents. As soon as the documents (signed informed consent, evaluation form, ERI, MBI, demographic questionnaire and the form for designation of the attending physician) are returned, the study manager contacts the employee and either tells him/ her that an appointment with the designated physician should be made within the following week (Neuropattern™ group) or that there will be a three months wait (control group). The employee attends the medical appointment with the designated physician and documents sent to the physician beforehand (NPQ-A, medical clearance form and prescription form for Dexamethasone) are completed. Upon return of these documents, the Neuropattern™ test kit (including the questionnaires NPQ-P, NPQ-PSQ, NPQ-S and PHQ as well as 16 Salivettes® for saliva sample collection, 0.25 mg Dexamethasone and a portable ECG device) is shipped to the subject and Neuropattern™ is conducted at home. After return of the test kit to DAaCRO, the subject is assigned to neuropattern and will gain access to individualized online counseling for three months. Evaluation (including an evaluation form, ERI and MBI) will take place at baseline as well as three and six months after onset of online counseling for assessment of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Employees aged 18 to 65 yrs
* fluent in written and spoken German
* medical clearance by their attending physician
* signed informed consent

Exclusion Criteria:

* known intolerance to steroids
* intake of steroids or benzodiazepines
* pregnancy or lactation
* any psychiatric diseases or current psychotherapy
* acute somatic illnesses, that currently require medical treatment
* obviously unsuited as subject (lack of cognitive or verbal skills)
* arrhythmia absoluta
* decision against the intake of Dexamethasone by physician or subject (e.g. known intolerance to steroids, personal or medical reasons)
* participation in any other study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Work incapacitation will be assessed through number of absent days and medical consultations in the past three months and items recording the ability to meet the demands at work. | at study inclusion as well as 3 and 6 months after Neuropattern™ stress diagnostics
  Within-subject differences in work incapacitation will be recorded at study inclusion as well as 3 and 6 months after Neuropattern™ stress diagnostics, between-subject differences in work incapacitation of the Neuropattern™ group and the control group will be assessed.

SECONDARY OUTCOMES:
quality of life | at study inclusion as well as 3 and 6 months after Neuropattern™ stress diagnostics
  Subjects' quality of life will be recorded at study inclusion as well as 3 and 6 months after Neuropattern™ stress diagnostics allowing changes to be assessed and the Neuropattern™ group will be compared to control group.
severity of symptoms | at study inclusion as well as 3 and 6 months after Neuropattern™ stress diagnostics
  The severity of symptoms will be recorded at study inclusion as well as 3 and 6 months after Neuropattern™ stress diagnostics. The Neuropattern™ group will be compared to the control group and changes within subjects over time will be analyzed.
scores in the Maslach Burnout Inventory (MBI) | at study inclusion as well as 3 and 6 months after Neuropattern™ stress diagnostics
  MBI scores will be recorded at study inclusion as well as 3 and 6 months after Neuropattern™ stress diagnostics. Changes within subjects will be analyzed and the Neuropattern™ group will be compared to the control group.
scores in the Effort-Reward Imbalance Questionnaire (ERI) | at study inclusion as well as 3 and 6 months after Neuropattern™ stress diagnostics
  ERI scores will be recorded at study inclusion as well as 3 and 6 months after Neuropattern™ stress diagnostics. Changes within subjects will be analyzed and the Neuropattern™ group will be compared to the control group.
exploring the frequency and combinations of neuropattern in a population with high demands at work | after the Neuropattern™ diagnosis is generated, approximately one month after study inclusion
  There are thirteen different neuropattern generated from biological psychological and symptomatic variables assessed by the Neuropattern™ questinnaires and the biomarkers. After the Neuropattern™ diagnosis is generated, approximately one month after study inclusion, frequency and combinations of neuropattern found in the study population will be documented as part of an evaluative and developmental process of Neuropattern™ stress diagnostics.

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Hellhammer, MSc, Principal Investigator — Daacro GmbH & Co. KG
Locations (1):
- DAaCRO GmbH & Co. KG, Trier, Rhineland-Palatinate, Germany

REFERENCES:
- [Background] Hellhammer, D. H., & Hellhammer, J. (2008). Stress- The Brain-Body Connection (Vol. 174). Basel: Karger.
- See also: DAaCRO homepage — http://www.daacro.de
- See also: Homepage of the University of Trier — http://www.uni-trier.de